CLINICAL TRIAL: NCT04325828
Title: An Open-label Phase 2 Study to Evaluate the Efficacy and Safety of Apalutamide in Combination With Gonadotropin-releasing Hormone (GnRH) Agonist in Subjects With Locally Advanced or Recurrent/Metastatic and Androgen Receptor (AR) Expressing Salivary Gland Carcinoma
Brief Title: A Study of Apalutamide Combined With GnRH Agonist in Participants With Androgen Receptor Positive Salivary Gland Carcinoma
Acronym: YATAGARASU
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108758; 56021927SGT2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Results first posted 2022-07-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Salivary Gland Neoplasms
MeSH Terms: conditions — Salivary Gland Neoplasms | interventions — apalutamide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Apalutamide plus GnRH Agonist (Experimental): Participants will receive apalutamide 240 milligram (mg) in combination with a gonadotropin-releasing hormone (GnRH) agonist until disease progression, unacceptable toxicity, death, or the end of the study and each treatment cycle will be of 28 days. Participants who are benefitting from this study will enter long term extension phase.
  Interventions: Drug: Apalutamide; Drug: GnRH Agonist

INTERVENTIONS:
Drug: Apalutamide — Apalutamide 240 mg (4*60-mg tablets) will be administered orally once daily with or without food.
  Other Names: JNJ-56021927
Drug: GnRH Agonist — A stable regimen of goserelin 3.6 mg will be administered as a GnRH agonist.

SUMMARY:
The purpose of the study is to evaluate the overall response rate (ORR) of apalutamide in combination with a gonadotropin-releasing hormone (GnRH) agonist in participants with androgen receptor (AR) expressing locally advanced or recurrent/metastatic salivary gland carcinoma (SGC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed salivary gland carcinoma (SGC) by local pathology
* Androgen receptor (AR) expressing SGC: Local testing of AR-positivity will be performed as standard of care for the eligibility confirmation. AR-positivity will be defined according to immunohistochemistry (IHC) staining of tumor tissue with at least 1 percent (%) of cell nuclei staining positive. Tissue should be available for the central confirmation of AR-positivity, but the central result of AR positivity will not be required for initiating the study intervention
* Locally advanced or recurrent/metastatic SGC
* Measurable lesion(s) according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2

Exclusion Criteria:

* Treatment with any other investigational agent or participation in another clinical study with therapeutic intent within 30 days prior to first dose. Treatment with a drug that has a short half life (t1/2) (for example, less than [<] 1 day) may be eligible in accordance with the discussion with the sponsor's medical monitor
* Radiographically confirmed brain metastases. In case of history of brain metastases that were previously treated and not recurred for at least 6 months, they are considered eligible
* Toxicities from previous anticancer therapies should have resolved to baseline levels or to Grade 1 or less (except for all grade alopecia, and for peripheral neuropathy, and hypothyroidism stable on hormone replacement therapy to be Grade 2 or less). If corticosteroids are administered for any reasons such as the management of toxicities due to prior therapies, the dose must be tapered until 10 milligram (mg)/day or less of prednisolone and contact the sponsor's medical monitor on an individual basis prior to the first dose
* Active or symptomatic viral hepatitis or chronic liver disease; ascites or bleeding disorders secondary to hepatic dysfunction
* History of seizure or any condition that may predispose to seizure (including, but not limited to, prior stroke, transient ischemic attack, or loss of consciousness less than or equal to [<=] 1 year prior to first dose; brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect)
* Treatment with drugs known to lower the seizure threshold within 4 weeks prior to first dose
* Known or suspected contraindications or hypersensitivity to apalutamide, gonadotropin-releasing hormone agonist (GnRHa) analogues or any of the components of the formulations
* Received prior ADT including a GnRH analogue, AR blocker such as bicalutamide, enzalutamide or 17alpha-hydroxylase-17,20-lyase (CYP17) inhibitor such as abiraterone acetate etc. Chemotherapy, radiation, or surgery as part of curative intent therapy are allowed so long as prior therapy did not include ADT. Prior chemotherapy, targeted cancer therapy or immunotherapy within 1 week or 4 half-lives whichever is longer, before the first administration of study drug. For agents with long half-lives, the maximum required time since last dose is 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2027-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (7):
- Japan (7):
  - National Cancer Center Hospital, Chūōku
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Kansai Medical University Hospital, Hirakata
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Aichi Cancer Center Hospital, Nagoya
  - Niigata University Medical And Dental Hospital, Niigata
  - Hokkaido University Hospital, Sapporo

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Apalutamide + Goserelin: Participants with androgen receptor (AR) expressing locally advanced or recurrent/metastatic salivary gland carcinoma (SGC) received apalutamide 240 milligrams (mg) (4*60 mg tablets) orally once daily with or without food in combination with stable regimen of goserelin 3.6 mg administered subcutaneously once per cycle (each cycle is of 28 days) as a gonadotropin-releasing hormone (GnRH) agonist, until disease progression, unacceptable toxicity, death, or end of the study.
Period: Overall Study
Arm/Group | Apalutamide + Goserelin
Started | 31
Completed | 5
Not Completed | 26
Not completed — Ongoing | 26

BASELINE CHARACTERISTICS:
Arm/Group | Apalutamide + Goserelin
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 65 [50 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 31
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR) was defined as the percentage of participants who achieve partial response (PR) or better according to the response evaluation criteria in solid tumors (RECIST) version1.1, including with either confirmed best overall response of complete response (CR) or PR during the study. CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeters (mm). PR is defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, in absence of new lesions or unequivocal progression of non-target lesions.
Time Frame: Up to 13 months
Population: Response evaluable set included all participants who were androgen receptor (AR) positive by local test and were confirmed evaluable by independent central radiology review (ICRR) and also, who received at least 1 dose of study drug and had at least 1 postbaseline disease assessment or died due to disease progression before first postbaseline disease assessment. Here, 'N' (number of participants analyzed) included 24 response evaluable participants who were analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Apalutamide + Goserelin
Number analyzed (Participants) | 24
percentage of participants | 25

2. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate (CBR) was defined as the percentage of participants who achieved a confirmed best overall response of CR, PR, or stable disease (SD) for at least 24 weeks based on RECIST version 1.1 during the study (and prior to subsequent therapy if any). CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, in absence of new lesions or unequivocal progression of non-target lesions. SD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 13 months
Population: Response evaluable set included all participants who were AR positive by local test and who were confirmed evaluable by an ICRR and also, all participants who received at least 1 dose of study intervention and who had at least 1 postbaseline disease assessment or died due to disease progression before the first postbaseline disease assessment. Here, 'N' (number of participants analyzed) included 24 response evaluable participants who were analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Apalutamide + Goserelin
Number analyzed (Participants) | 24
percentage of participants | 50

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who achieved a confirmed best overall response of CR, PR, or SD based on RECIST version 1.1 during the study (and prior to subsequent therapy if any). CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, in absence of new lesions or unequivocal progression of non-target lesions. SD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 13 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Apalutamide + Goserelin
Number analyzed (Participants) | 24
percentage of participants | 70.8

4. Secondary Outcome: Progression-free Survival (PFS) as Assessed by ICRR
Description: PFS was defined as the time from the date of the initial dose of study intervention to the date of first documented disease progression as defined in the RECIST version 1.1, or death due to any cause, whichever occurred first. Progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: Up to 13 months
Population: Treated analysis set included all participants who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Apalutamide + Goserelin
Number analyzed (Participants) | 31
months | 7.43 [3.65 to NA] — The upper limit of 95% confidence interval was not estimable due to less number of participants with events.

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from the date of the initial dose of study intervention to the date of the participant's death.
Time Frame: Up to 13 months
Population: Treated analysis set included all participants who received at least 1 dose of study intervention.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Apalutamide + Goserelin
Number analyzed (Participants) | 31
months | NA [NA to NA] — The median and 95% confidence interval were not estimable due to very less number of participants with events.

6. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined among responders (with a CR or PR) as the time between date of the initial dose of study intervention and the first efficacy evaluation that the participant had met all criteria for CR or PR. CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, in absence of new lesions or unequivocal progression of non-target lesions.
Time Frame: Up to 13 months
Population: Population analyzed included response evaluable set amongst who were responders (CR or PR).
Measure: Median (Full Range); unit: months
Arm/Group | Apalutamide + Goserelin
Number analyzed (Participants) | 6
months | 1.87 [1.7 to 3.7]

7. Secondary Outcome: Duration of Response (DoR)
Description: DoR calculated among responders from the date of initial documentation of a response (CR or PR) to the date of first documented evidence of progressive disease as defined in RECIST version 1.1 or death, whichever occurred first. CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is defined as at least a 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters, in absence of new lesions or unequivocal progression of non-target lesions.
Time Frame: Up to 13 months
Population: Population analyzed included response evaluable set amongst who were responders (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Apalutamide + Goserelin
Number analyzed (Participants) | 6
months | NA [6.64 to NA] — The median and upper limit of 95% confidence interval were not estimable due to very less number of participants with events.

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs were reported. Treatment-emergent adverse events (TEAEs) for the treatment phase included events with an onset date/time on or after the start of study intervention through the day of last dose plus 30 days were considered as treatment-emergent.
Time Frame: Up to 13 months
Population: Safety analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Apalutamide + Goserelin
Number analyzed (Participants) | 31
Participants | 28

9. Secondary Outcome: Plasma Concentration of Apalutamide
Description: Plasma concentration of apalutamide was reported.
Time Frame: Day 1 (predose) of Cycles 2 to 6 (each cycle was of 28 days)
Population: Pharmacokinetics analysis set included all participants with at least 1 apalutamide and/or N-desmethyl apalutamide concentration data after the first study intervention administration. Here, 'N' (number of participants analyzed) specifies all participants who were evaluated for this outcome measure (OM). Here, 'n' (number analyzed) specifies the number of participants evaluated at specified timepoints.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | Apalutamide + Goserelin
Number analyzed (Participants) | 29
micrograms per milliliter (mcg/mL)
  Cycle 02 Day 1, Predose | 4.67 (1.19)
  Cycle 03 Day 1, Predose: number analyzed (Participants) | 28
  Cycle 03 Day 1, Predose | 4.32 (1.35)
  Cycle 04 Day 1, Predose: number analyzed (Participants) | 25
  Cycle 04 Day 1, Predose | 4.05 (1.46)
  Cycle 05 Day 1, Predose: number analyzed (Participants) | 23
  Cycle 05 Day 1, Predose | 4.18 (1.38)
  Cycle 06 Day 1, Predose: number analyzed (Participants) | 19
  Cycle 06 Day 1, Predose | 4.16 (1.52)

10. Secondary Outcome: Plasma Concentration of N-desmethyl Apalutamide
Description: Plasma concentration of N-desmethyl Apalutamide was reported.
Time Frame: Day 1 (predose) of Cycles 2 to 6 (each cycle was of 28 days)
Population: Pharmacokinetics analysis set included all participants with at least 1 apalutamide and/or N-desmethyl apalutamide concentration data after the first study intervention administration. Here, 'N' (number of participants analyzed) specifies all participants who were evaluated for this OM. Here, 'n' (number analyzed) specifies the number of participants evaluated at specified timepoints.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Apalutamide + Goserelin
Number analyzed (Participants) | 29
mcg/mL
  Cycle 02 Day 1, Predose | 7.19 (1.21)
  Cycle 03 Day 1, Predose: number analyzed (Participants) | 28
  Cycle 03 Day 1, Predose | 6.89 (1.56)
  Cycle 04 Day 1, Predose: number analyzed (Participants) | 25
  Cycle 04 Day 1, Predose | 6.29 (1.66)
  Cycle 05 Day 1, Predose: number analyzed (Participants) | 23
  Cycle 05 Day 1, Predose | 6.53 (1.81)
  Cycle 06 Day 1, Predose: number analyzed (Participants) | 19
  Cycle 06 Day 1, Predose | 6.40 (1.91)

ADVERSE EVENTS:
Time Frame: Up to 13 months
Description: Safety analysis set included all participants who received at least 1 dose of study intervention.
Arm/Group | Apalutamide + Goserelin
All-Cause Mortality (participants affected / at risk) | 4/31
Serious Adverse Events (participants affected / at risk) | 5/31
Other Adverse Events (participants affected / at risk) | 28/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apalutamide + Goserelin (N=31)
Anaemia (Blood and lymphatic system disorders) | 1
Oesophageal Stenosis (Gastrointestinal disorders) | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cerebral Infarction (Nervous system disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apalutamide + Goserelin (N=31)
Anaemia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 2
Hypothyroidism (Endocrine disorders) | 6
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 2
Malaise (General disorders) | 5
Upper Respiratory Tract Infection (Infections and infestations) | 2
Radiation Skin Injury (Injury, poisoning and procedural complications) | 2
Blood Creatinine Increased (Investigations) | 2
Blood Thyroid Stimulating Hormone Increased (Investigations) | 3
Weight Decreased (Investigations) | 4
Decreased Appetite (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 8
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 10
Hot Flush (Vascular disorders) | 6
Hypotension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
Due to the low numbers of female participants, it was difficult to interpret the difference between males and females. There was a lack of data on individual treatment of apalutamide as well as goserelin. The number of participants in this study was limited, and the follow-up period was immature at this cut-off for the primary analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT04325828/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT04325828/SAP_001.pdf